CLINICAL TRIAL: NCT07278778
Title: A Pilot Study of Cancer Care Companion, An Electronic Health Record Tool to Improve Information Exchange and Self-Management in Pediatric Cancer
Brief Title: Cancer Care Companion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 202601022; 1R21CA290223-01A1 (NIH)
Record Dates: First submitted 2025-12-05; First posted 2025-12-12 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Cancer
Keywords: communication; electronic medical record; pediatric cancer
MeSH Terms: conditions — Neoplasms; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Participants (Experimental): All participants receive the Cancer Care Companion program. There is no control or comparison group.
  Interventions: Other: Cancer Care Companion

INTERVENTIONS:
Other: Cancer Care Companion — The investigators will provide parents access the Cancer Care Companion through Epic MyChart. If a participant has not enrolled in MyChart, the investigator will provide instructional materials and assist with registration. Parents will use the Cancer Care Companion for 3 months during which they will complete tasks including educational modules, check-in surveys, and patient stories. Participants may opt-out of receiving the patient stories. During the 3-month intervention, participants will receive 13 educational tasks, 7 check-in surveys, and 5 patient stories (if requested). The Day 1 educational task will include an overview of the program and further instructions. After enrollment, participants will retain access to Cancer Care Companion for at least 3 months, during which they can revisit the content.

SUMMARY:
This study invites parents of children with cancer to use an electronic health record (EHR)-based communication tool, called the Cancer Care Companion, and assess the acceptability, appropriateness, and feasibility of the tool.

DETAILED DESCRIPTION:
High-quality communication between clinicians and parents is critical to providing optimal care for pediatric cancer. This study engages parents of children with cancer to use an electronic health record (EHR)-based communication tool, called the Cancer Care Companion, and assess the acceptability, appropriateness, and feasibility of the tool. Parent participants will be given 3 months of access to Cancer Care Companion, after which the participant(s) will complete a semi-structured interview. Participants will also complete a survey of validated measures before and after the intervention.

ELIGIBILITY:
Eligibility Criteria for Parents:

Parents of children with cancer will be enrolled if they meet the following criteria:

* They are a legal guardian of a child diagnosed with cancer in the prior 4 weeks.
* The child plans to receive or currently receives cancer directed therapy at St. Louis Children's Hospital.
* The parent or legal guardian has access to internet through a computer or smart phone.
* Speaks and reads in English
* The parent or legal guardian agrees to enroll in Epic MyChart to access a proxy portal for their child.

Eligibility Criteria for Clinicians:

* Clinicians with patients who have parents participating may be enrolled. Clinician participants will be employed at SLCH or Washington University School of Medicine (WUSM). The clinicians will include physicians, nurse practitioners, and nurse coordinators from the leukemia/lymphoma, brain tumor, and solid tumor teams in order to represent the breadth of pediatric cancer diagnoses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-04 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Tool feasibility | Immediately post-intervention
  The number of tasks marked "complete" divided by total tasks delivered, reported as a percentage per participant, with success defined as meeting or exceeding a 70% completion rate.

SECONDARY OUTCOMES:
Information Exchange | Baseline and immediately post-intervention
  Health Literacy of Caregivers Scale-Cancer is a validated tool measuring 10 domains relevant to caregiver health literacy. The information exchange domain includes 4 items with a 4-point Likert response scale assessing whether caregivers have adequate information about cancer and cancer management.
Trust in Physicians | Baseline and immediately post-intervention
  The Trust in Physician Scale is an 11-item tool using a 5-point Likert response scale to assess respondents' perceptions of their doctors' ability to manage (diagnose, treat, make appropriate referrals) their health problem.
Ability to navigate the healthcare system | Baseline and immediately post-intervention
  Health Literacy of Caregivers Scale-Cancer is a validated tool measuring 10 domains relevant to caregiver health literacy. The healthcare system domain includes 6 items with a 4-point Likert response scale assessing whether caregivers understand the healthcare system and how to find care for their child.
Caregiver burden | Baseline and immediately post-intervention
  The short version of the Burden Scale for Family Caregivers is a validated 10-item tool with a 4-point Likert response scale assessing caregiver burden and how it affects the caregivers' physical, mental, and social well-being.
Parental anxiety | Baseline and immediately post-intervention
  The PROMIS Anxiety SF 4a is a validated 4-item tool with a 5-point Likert response scale used to measure emotional distress and anxiety.
Communication Quality | Baseline and immediately post-intervention
  The PedCOM Short Form is a validated 8-item tool using a 5-point Likert response scale that assesses dimensions of communication quality (information exchange, building relationships, making decisions, responding to emotions, supporting hope, providing validation, managing uncertainty, and enabling self-management).
Patient perceptions of tool usability | Immediately post-intervention
  The System Usability Scale is a validated 10-item tool with a 5-point Likert response scale that measures users perceptions of the complexity, usability, functionality, and value of technological systems.
Patient perceptions of tool usefulness | Immediately post-intervention
  The semi-structured interview guide will be developed using the Unified Theory of Acceptance and Use of Technology and theory of Technology Readiness.
Patient perceptions of tool barriers and facilitators | Immediately post-intervention
  The semi-structured interview guide will be developed using the Unified Theory of Acceptance and Use of Technology and theory of Technology Readiness.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan A Sisk, MD, MSCI, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine/Saint Louis Children's Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be submitted to the Qualitative Data Repository at Syracuse University.
Supporting Information: Study Protocol, ICF

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu